CLINICAL TRIAL: NCT02051361
Title: Open Label, Non Interventional, Multi-center, Observational Study to Assess the Antiplatelet Treatment Pre and Post-operatively of Stent Implantation
Brief Title: Antiplatelet Therapy Following Stent Implantation
Acronym: Anti-Clot
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-CLOBES-EL-41
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Acute Myocardial Infarction; Coronary Syndrome; Angina, Unstable
Keywords: DAT = Dual Antiplatelet Treatment; Major Cardiac Adverse Events
MeSH Terms: conditions — Angina, Unstable; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clopidogrel treated patients: Patients pre and post operatively following stent implantation treated with clopidogrel and aspirin

SUMMARY:
Coronary artery stents, particularly drug-eluting stents (DES), are used in the majority of patients who undergo percutaneous coronary intervention (PCI) to improve symptoms in patients with obstructive coronary artery disease. They function both to prevent abrupt closure of the stented artery soon after the procedure as well as to lower the need for repeat revascularization compared to balloon angioplasty alone . Stent restenosis and stent thrombosis are potential complications of coronary artery stenting; their incidence is highest in the first year after PCI. Stent restenosis, which occurs more frequently with bare metal stents (BMS) than DES, may occasionally present as an acute myocardial infarction (MI). Stent thrombosis is an uncommon but serious complication that often presents as death and is almost always accompanied by MI, usually with ST-segment elevation. Patients are commonly treated with dual antiplatelet therapy (DAPT) for the recommended duration for the particular stent. DAPT (aspirin plus platelet P2Y12 receptor blocker) and significantly lowers the risk of stent thrombosis.

DETAILED DESCRIPTION:
New Guidance on Antiplatelet Therapy After Stenting: Clinical Advisory, Kirsten E. Fleischmann, MD, MPH reviewing Grines CL et al. Circulation 2007 Feb 13. An expert panel recommends 12 months of therapy after placement of drug-eluting stents. Aspirin and clopidogrel are commonly prescribed after placement of both bare metal stents and drug-eluting stents. However, recent concerns about stent thrombosis (Journal Watch Jan 4 2007) have led experts from multiple groups, including the American Heart Association and the American College of Cardiology, to issue an advisory on preventing premature discontinuation of dual antiplatelet therapy. Based on a review of the literature, the experts offer observations and recommendations including the following:

* Dual antiplatelet therapy with aspirin and a thienopyridine such as clopidogrel reduces cardiac events after coronary stenting.
* Premature discontinuation of these agents greatly increases the risk for stent thrombosis and associated clinical events such as myocardial infarction and death.
* Patients should receive 12 months of dual antiplatelet therapy after placement of drug-eluting stents.
* Elective surgery associated with a significant risk for bleeding should be postponed until an appropriate course of dual antiplatelet therapy (i.e., 1 month for bare metal stents and 12 months for drug-eluting stents) has been completed.
* Patients' ability to comply with prolonged dual antiplatelet therapy and their need for subsequent invasive procedures should be considered when choosing the type of stent.
* Patients and their other providers should consult with the patient's cardiologist before stopping dual therapy.

Endpoints:

Primary endpoint - Outcome Measures:

1. Major Cardiovascular events at 1, 3, 6, 12 months after study enrolment

* All Death,
* Cardiac death,
* Myocardial infarction,
* Stroke,
* Target vessel revascularization
* Bleeding event
* In-stent restenosis (ISR)

  * Angiographical Determination of Binary Stenosis Rate (defined as diameter stenosis of at least 50 % in the stent and / or persistent area, 6, 9, 12 months after stent implantation) The angiographical determination of the degree of stenosis, defined as percentage diameter stenosis in the stent and /or persistent area, 6 and 12 months after stent implantation.
  * The angiographical determination of the minimal lumen diameter in the stent and / or persistent area, 6 months after stent implantation.

Secondary:

* Description of any reported AE/ SAE per study subgroup.
* Description of any missing doses per study subgroup.

Study Medication:

Category: ADP-P2Y12 interaction blokers

* Clopidogrel (Clovelen®)
* Dosage: As per Clopidogrel (Clovelen®) SmPC

Study Concomitant Medication:

Aspirin. DAT = Dual antiplatelet therapy consists of aspirin add on clopidogrel

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom planned or unplanned stent implantation
* Ages Eligible for Study: 18 Years and older
* Genders Eligible for Study: Both
* Acute coronary syndrome
* ST-segment elevation MI (STEMI)
* non ST-segment elevation MI (STEMI)
* Stable angina pectoris and or/ documented myocardial ischemia
* Instable angina pectoris and or/ documented myocardial ischemia
* De-novo stenosis of coronary artery with a degree of stenosis between 50% and 99%, that is accessible to PTCA
* Patients on pre-defined group of clopidogrel treatment during and after DES implantation
* Willingness and ability to adhere to the study conditions
* Written informed consent after patient information

Exclusion Criteria:

* Known severe arrhythmias that necessitate a long term antiarrhythmic therapy
* Pericarditis
* Intracardiac thrombus
* Bacterial endocarditis
* Patients with contraindication for aortocoronary bypass operation,
* Contraindication to antiplatelet therapy
* Non-cardiac co-morbid conditions that may result in protocol non-compliance (per site investigator's medical judgment).
* Bleeding diathesis
* Thrombocytopenia (<150 000/mm3)
* Recent (<6 months) gastrointestinal bleeding
* Recent stroke within 6-months
* Concurrent organ damage (creatinine level > 2.0mg/dL or AST and ALT > 3 times upper normal reference values)
* Patients with left main stem stenosis (>50% by visual estimate)
* History of allergy to aspirin
* Inability, to understand sense and purpose of the study
* Patients not willing to keep the conditions of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on clopidogrel treatment following stent implantation
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of Major Adverse Cardiac Events (MACEs) | 6 months
  All Death,
  * Cardiac death,
  * Myocardial infarction,
  * Stroke,
  * Target vessel revascularization (TVR)
  * Bleeding event
  * In-stent restenosis (ISR)

SECONDARY OUTCOMES:
Number of missed daily doses | 6 months
  Compliance to antiplatelet treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Patsilinakos, MD, PhD, Study Director — Agia Olga Konstantopoulion hospital of Athens; Nikolaos Kafkas, MD Cardiologist, Principal Investigator — KAT Hospital of Athens
Locations (1):
- KAT Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://circ.ahajournals.org/content/117/2/261.full.pdf
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/17224480
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19044176
- See also: Related Info — http://www.ima.org.il/FilesUpload/IMAJ/0/43/21642.pdf
- See also: Related Info — http://www.scielo.br/pdf/jvb/v7n3/v7n3a10.pdf